CLINICAL TRIAL: NCT01887353
Title: A Randomized, Double-blind, Placebo Controlled Study, Designed to Investigate the Effect of Ranolazine on Left Ventricular Diastolic Function in Patients With Symptomatic AF and Preserved Ejection Function, After the Subject Has Undergone a Successful External Electrical Cardioversion
Brief Title: The Use of Ranolazine for Atrial Fibrillation and Diastolic Heart Failure
Acronym: RAD HF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficultly in enrolling
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1024475
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: atrial fibrillation; heart failure; ranolazine; cardioversion; persistent AF; paroxysmal AF
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator)
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Patients will take ranolazine 1000 mg tablets twice daily
  Arms: Ranolazine
Drug: Placebo — Placebo pill manufactured to mimic ranolazine 1000 mg tablets. Patients will be instructed to take two pills a day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of ranolazine in the prevention of recurrent atrial fibrillation in post-cardioversion patients with heart failure and preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female > 18 years of age;
* Documentation of heart failure and who are in NYHA class II or III;
* Documented history of symptomatic AF < 6 months in duration at the time of presentation, currently in AF at the time of the external electrical cardioversion, and successfully restored to normal sinus rhythm;
* Percutaneous coronary intervention (PCI) patients who can be placed on anticoagulation with warfarin post-cardioversion (and not on rivaroxaban or dabigatran);
* Demonstration of preserved ejection fraction (EF) by echocardiography;
* Echocardiographic evidence of impaired diastolic filling.

Exclusion Criteria:

* Known history of permanent or long-standing AF (> 6 months);
* Other acutely reversible causes of AF, including but not limited to: hyperthyroidism, pericarditis, myocarditis or pulmonary embolism;
* Known history of cirrhosis;
* NYHA Class IV;
* Myocardial Infarction, unstable angina, or coronary artery bypass graft surgery within three months prior to screening;
* Percutaneous coronary intervention (PCI) within 4 weeks prior to screening, if these patients need to be placed on rivaroxaban or dabigatran post-cardioversion;
* Clinically significant valvular disease;
* Clinically significant pulmonary disease;
* Stroke within 3 months prior to screening;
* Creatinine clearance < 30 mL/min as calculated by Cockcroft-Gault formula;
* Use of anti-arrhythmic drugs (Class Ia or IIIc) within 3 months prior to screening;
* Concurrent use of drugs considered strong inhibitors of CYP3A;
* Concurrent use of drugs considered as CYP3A inducers;
* Prior treatment with ranolazine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T. Jared Bunch, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 4 | 4
Completed | 0 (Study was stopped early because of difficulty recruiting.) | 1 (Study was stopped early because of difficulty recruiting.)
Not Completed | 4 | 3
Not completed — Study stopped early | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 89.7 (9.5) | 78.9 (8.9) | 84.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to First Atrial Fibrillation (AF) Recurrence
Description: There were too few participants for an assessment of time to first recurrence, therefore the numbers of participants with recurrence up to 6 months is reported instead
Time Frame: up to 6 months
Measure: Number; unit: participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 4 | 4
participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Entire study duration (up to 6 months or until stoppage).
Arm/Group | Ranolazine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=4) | Placebo (N=4)
Medication intolerance (Cardiac disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes